Oral combined Hydrochlorothiazide/Lisinopril versus oral nifedipine for postpartum hypertension: A comparative effectiveness pilot randomized

NCT05049616

Version Date: 07/06/2022

Oral combined Hydrochlorothiazide/Lisinopril versus oral nifedipine for postpartum hypertension: A comparative effectiveness pilot randomized controlled trial

**Study protocol** 

Principal investigator: Michal Fishel Bartal, MD

Co-investigators:

Baha Sibai, MD

Sean Blackwell, MD

Joyce P. Samuel, MD

Division of Maternal-Fetal Medicine, Department of Obstetrics, Gynecology and Reproductive Sciences, The University of Texas Health Science Center at Houston

## **Background and significance:**

Hypertensive disorders of pregnancy (HDP) complicate up to 10% of pregnancies and are a significant cause of maternal mortality and morbidity.1 Hypertension may be present before or during pregnancy or in postpartum. Postpartum hypertension can be related to the persistence of gestational hypertension, preeclampsia, preexisting chronic hypertension, or it could develop de novo secondary to other causes. While most research efforts have mainly been focused on the antenatal management of hypertension for a maternal and fetal benefit, there is a paucity of studies evaluating the behavior of postpartum hypertension and the pharmacologic therapies during this period to optimize maternal safety and minimize hospital stay.

Postpartum hypertension results in increased medical costs due to prolonged hospitalization, the need for magnesium sulfate and antihypertensive drugs, and increased hospital readmission rates. People with hypertensive disorder of pregnancy are at increased risk for immediate postpartum complications, including hypertensionrelated complications (i.e., uncontrolled blood pressure, acute cardiovascular disease, acute cerebrovascular disease, acute renal insufficiency), and obstetric related postpartum complications (i.e., infection, hemorrhage, venous thromboembolism). <sup>2</sup> Hypertensive disorder of pregnancy, and chronic hypertension are a risk factor for stroke during the postpartum period, with the majority of stroke readmission after birth occurring in the first 10 days after discharge. <sup>3</sup> Despite the cure for preeclampsia being the delivery of the infant, maternal health implications persist well beyond the pregnancy. Preeclampsia is associated with maternal cardiovascular dysfunction and

long-term cardiovascular risk,<sup>4-9</sup> including a 2-fold risk of ischemic heart disease and stroke and a 4-fold risk of hypertension in later life.<sup>7,8,10-12</sup> The association between preeclampsia and future CVD persists, despite accounting for mutual risk factors, including age, obesity, and prepregnancy hypertension.<sup>13</sup> Cardiovascular disease is not only more common in people with preeclampsia, but it tends to occur earlier, with a higher fatality rate. <sup>8</sup>

For many asymptomatic women, antenatal care is their first adult engagement with the healthcare system. Consequently, pregnancy and the early postpartum provide an ideal window for risk screening and primary prevention of long-term cardiovascular health and future pregnancy outcomes.

The American College of Obstetricians and Gynecologists (ACOG) recommends close outpatient blood pressure monitoring in all women with preeclampsia 7-10 days (or sooner if the patient is symptomatic) after delivery as the standard of care. Blood pressure rises progressively over the first five postnatal days, peaking on days three to six after delivery.

## Blood pressure medication during the postpartum period:

During the immediate hospital stay after delivery, antihypertensive medications are recommended after delivery if systolic BP remains persistently ≥150 mm Hg and/or if diastolic BP ≥ 100 mm Hg. <sup>14</sup> However, there are no clear guidelines on optimal blood pressure management in the postpartum period. Based on previous data, at least 60-70% of women diagnosed with preeclampsia before delivery will require BP medications at discharge. <sup>15-17</sup> <sup>18</sup>At three months postpartum, 39% of women still had hypertension



(defined as blood pressure ≥140/90), which decreased to 18% at two years postpartum.

17

A case-control study has also found that readmitted patients with HDP were less likely to start antihypertensive medications during their initial hospitalization after controlling for age, race, and chronic hypertension. <sup>19</sup> Based on previous data during readmission for hypertension, more than 50% of patients will start hypertensive medications. <sup>20</sup>

Despite the widespread use of antihypertensive drugs in the postpartum period, there is limited evidence regarding the preferred antihypertensive agent in that period (Table1). Usually, the selection of the antihypertensive agent is based on clinical judgment, as there are no standardized management guidelines for specific antihypertensive agents or parameters for postpartum medication titration.<sup>18</sup>

Table 1: Randomized controlled studies evaluating medications for postpartum hypertension

| Study/<br>Year | n/<br>Total<br>number of<br>patients | Intervention | Control | Primary<br>outcome | Results |
|---|---|---|---|---|---|
| Calcium ch | nannel blocke | ers | | | |
| Barton <sup>21</sup> /<br>1990 | Severe<br>preeclamp<br>sia<br>N=32 | Nifedipine<br>(oral,10mg) | Placebo | MAP | Reduction in<br>MAP with<br>nifedipine<br>between 18-<br>24 hours<br>postpartum<br>(93.9 versus<br>100.2 mm<br>Hg; p less<br>than 0.05) |

| Vermillion <sup>22</sup> /1998 | Severe BP<br>(170/105)<br>N=50 | Nifedipine<br>(oral,10mg) | Labetalol<br>20mg IV | Time to<br>achieve<br>therapeutic<br>goal<br>(<160/100) | Time to<br>achieve BP<br>goal shorter<br>with<br>nifedipine<br>(25 ± 13.6<br>min vs. 43.6<br>±25.4 min; P<br>=.002). |
|---|---|---|---|---|---|
| Arias-<br>Hernande<br>z <sup>23</sup> /2020 | Postpartu<br>m<br>preeclamp<br>sia with<br>severe<br>features<br>N=42 | Diltiazem<br>(oral,60mg TID) | Nifedipin<br>e<br>(oral,10m<br>g TID) | SBP, DBP,<br>MAP | At 6 hours, lower SBP (133.4±10.2) vs. 147.9 ±9.7,p<0.00 1) and DBP (78.5±7.7) vs. 90.6 ±5.5, p<0.001) with Diltiazem |
| Beta-block | er | | | | |
| Fidler <sup>24</sup> /<br>1982 | Postpartu<br>m HTN<br>(DBP 95-<br>105)<br>N=80 | Timolol (oral) | Methyldo<br>pa (oral) | SBP, DBP | Lower SBP<br>with Timolol<br>(difference<br>5.1mmHg,<br>p<0.05) |
| Mabie <sup>25</sup> /<br>1987 | Severe<br>Postpartu<br>m HTN<br>(DBP>110)<br>N=60 | Labetalol (IV 20-<br>80mg) | Hydralazi<br>ne (IV<br>5mg) | MAP | Improved in<br>the control<br>group<br>(difference<br>5.1mmHg,<br>p<0.02) |
| Sharma <sup>26</sup> /<br>2017 | Postpartu<br>m HTN<br>(>150/100)<br>N=50 | Labetalol (oral<br>200mg BID) | Nifedipin<br>e (30mg<br>daily) | Time to BP control | No<br>difference<br>(37.6 hours<br>versus 38.2<br>hours, p =<br>0.51) |
| Diuretics | Γ = | T = | 1 = : | T = - | |
| Matthews <sup>2</sup> <sup>7</sup> /1997 | Preeclamp<br>sia<br>N=19 | Furosemide (oral,<br>40mg, 7 days) | Placebo | Mean BP,<br>Max BP | No<br>difference |
| Ascarelli <sup>28</sup><br>/2005 | Preeclamp<br>sia<br>N=264 | Furosemide (oral, 20mg, 5 days) + | Placebo | SBP | No benefit<br>for patients<br>with mild |



| | | Oral potassium supplementation | | | preeclampsi a (n = 169) or superimpose d preeclampsi a (n = 25). Patients with severe preeclampsi a had lower SBP (142±13 mm Hg vs 153±19 mmHg, P < .004), and required less antihyperten sive therapy during hospitalizatio n (14% vs 26%, P = .371) |
|---|---|---|---|---|---|
| Venna <sup>29</sup> /<br>2017 | Postpartu<br>m HTN<br>(>150/100)<br>N=108 | Furosemide (oral,<br>20mg, 3 days) +<br>Nifedipine (10mg<br>TID) | Nifedipin<br>e (10mg<br>TID) | SBP,DBP,<br>MBP, need<br>for<br>additional<br>HTN drugs | No difference in BP. Requirement of additional antihyperten sive higher in in Nifedipine alone group (26.0% vs. 8.0%, p = 0.017) |
| Viteri <sup>30</sup> /<br>2018 | Preeclamp<br>sia<br>N=118 | Torsemide (20<br>mg, 5 days) | Placebo | BP>150/10<br>0 by day 5<br>or<br>discharge | No<br>difference |
| Perdigao <sup>3</sup> 1/ 2021 | Gestational<br>hypertensi<br>on/preecla<br>mpsia | Furosemide (oral,<br>20mg, 5 days) | Placebo | persistent<br>hypertensi<br>on 7 days<br>postpartum | 60% reduction in the prevalence |



| | N= 384 | | | (at least 2 consecutive BP readings over 48 hours of SBP ≥140 and DBP ≥90) | of persistent<br>hypertension<br>at 7 days<br>(adjusted<br>relative risk,<br>0.40 [95%<br>CI, 0.20–<br>0.81]) |
|---|---|---|---|---|---|
| ACE inhibi | | | | | |
| Ormesher <sup>32</sup> /2020 | Preterm<br>preeclamp<br>sia<br>N= 60 | Enalapril 5 mg daily for 1 week> 10 mg for 2 weeks then 20 mg maintenance dose for 6 month | Placebo | reduction in total vascular resistance from baseline to 6 months | No<br>difference |
| Alpha agoi | nists | | | | |
| Carlos<br>Noronha<br>Neto <sup>33</sup> /<br>2017 | Severe<br>HTN<br>(≥180/110)<br>N=90 | Clonidine (oral,<br>0.1mg) | Captopril<br>(oral,<br>25mg) | frequency<br>of very<br>high BP<br>episodes<br>(≥180/110)<br>while in the<br>obstetric<br>ICU | No<br>difference |
| Hydralazin | | | | | |
| Griffis <sup>34</sup> /<br>1989 | Gestational<br>HTN<br>N=26 | Hydralazine | Methyldo<br>pa | MAP | No<br>difference |
| Vigil-De<br>Gracia <sup>35</sup> /<br>2007 | Severe<br>HTN<br>(≥160/110)<br>N=82 | Hydralazine (IV,<br>5mg) | Labetalol<br>(IV,<br>20mg) | Persistent<br>severe BP | No<br>difference |

SBP; systolic blood pressure, DBP; diastolic blood pressure, MAP; mean arterial pressure

Angiotensin-converting enzyme inhibitors (ACE inhibitors) in the postpartum period.

A review of the available observational literature concluded that the following drugs have minimal milk to maternal plasma ratios to make breastfeeding acceptable: methyldopa, beta-blockers with high protein binding, angiotensin-converting enzyme inhibitors, and some dihydropyridine calcium channel blockers. <sup>36</sup> These drugs are used in the postpartum period, but the most common hypertensive treatment for antepartum and postpartum hypertension is Nifedipine and Labetalol. <sup>37</sup> ACE inhibitors are not used during pregnancy due to the higher risk for teratogenic effects but may be used in the postpartum period. ACE inhibitors are recommended for those with pregestational diabetes mellitus or cardiomyopathy and are the 1st drug of choice by the National Institute for Health and Care Excellence (United Kingdom) for postpartum hypertension. <sup>37-39</sup>

ACE inhibitors play an important role in controlling blood pressure outside of pregnancy. There is extensive evidence to support their cardioprotective effects. The HOPE (Heart Outcomes Prevention Evaluation) study, during which participants at high risk of cardiovascular disease were randomized to ramipril or placebo, was stopped prematurely due to the 22% reduction in myocardial infarction, cerebrovascular accident, or death from cardiovascular disease.<sup>40</sup>

ACE inhibitors may be used in the postpartum period without effect on breastfeeding, but the evidence on the effect of ACE inhibitors on postpartum hypertension treatment is limited.<sup>32,38,41-44</sup>

Normal pregnancy has been identified as a state of relative resistance to the pressor effects of Angiotensin II (Ang II).<sup>45</sup> In contrast, pregnant people with new-onset hypertension demonstrate increased sensitivity to the pressor effects of Ang II, even before the onset of hypertension.<sup>45,46</sup> Increased sensitivity to angiotensin II observed during pregnancy in women with hypertensive pregnancy was also present postpartum.<sup>47</sup> There is only one randomized study comparing captopril and clonidine for severe range blood pressure in the postpartum period. The above study concluded that both clonidine and captopril were safe and effective treatments for severe postpartum hypertension.<sup>33</sup> There are no studies to date comparing ACE inhibitors to other oral medications to control non-severe blood pressure in the postpartum period.

A recent randomized, double-blind placebo-controlled trial evaluated six months' treatment with enalapril to improve postnatal cardiovascular function in women with preterm preeclampsia. The primary clinical outcome was reduction in total vascular resistance (TVR) from baseline to 6 months post randomization following treatment with enalapril, compared with placebo. There was no difference in the TVR between groups at 6 months postpartum. Similarly, there was no difference in systolic function (measured by left ventricular ejection fraction/global longitudinal strain). However, individuals who were treated with enalaprilhad a significantly better diastolic function and improved LV remodeling, compared with placebo at 6 months than those treated with placebo. 32

Our experience with ACE inhibitors in the postpartum period has been favorable, but given the lack of data regarding use of ACE inhibitors in the postpartum period, it may not be an adequate drug for first-line treatment for persistent postpartum hypertension.

Diuretic use in the postpartum:

In individuals with preeclampsia, persistent hypertension and edema result in part from

the mobilization of up to 8 liters of fluid and sodium from the extravascular to

intravascular space. The increased urinary sodium excretion on days 3-5 postpartum

likely results from higher atrial natriuretic peptide concentrations in plasma and

activation of the renin-angiotensin-aldosterone system. Adding diuretics for postpartum

hypertension has been associated with better blood pressure control in some of the

studies.28,29

Rationale for a Clinical Trial and Hypothesis

CVD is the leading cause for mortality worldwide.

Primary prevention is more effective than treating CVD.

o Pregnancy is often the 1st adult engagement with the healthcare system.

o Preeclampsia is a risk factor for long term CVD, even after controlling for mutual

risk factors.

CVD is the leading cause for pregnancy related mortality.

There is no good data regarding the optimal medications to control blood

pressure after delivery.

ACE inhibitors play an important role in controlling blood pressure outside of

pregnancy and there is extensive evidence to support their cardioprotective

effects.

The optimal use of diuretics in the postpartum in patients with preeclampsia,

require further study and clarification to augment current management schemes.

UTHealth The University of Texas

**Hypothesis:** We hypothesize that in postpartum women with hypertensive disorders,

oral combined Hydrochlorothiazide/Lisinopril will reduce postpartum hypertension at 7

days after delivery compared to usual care with calcium channel blockers.

**PICO** question:

**Population:** Puerperal women with hypertension within the first 72 hours after delivery.

**Intervention:** Hctz/Lisinopril for postpartum management of hypertension

Comparison: Extended release nifedipine

Outcome: Stage 2 hypertension at day 7-10 after delivery (defined as SBP ≥ 140

and/or DBP ≥ 90 mmHg) or admission to the hospital for blood pressure control prior to

day 10.

Inclusion Criteria

Postpartum women at ≥ 18 years of age

Postpartum diagnosis of persistent hypertension (2 measurements of Systolic BP

≥150 and/or diastolic BP ≥ 100 or systolic BP ≥140 and/or diastolic BP ≥ 90 for

people with diabetes) requiring an oral medication based on the ACOG criteria or

Hypertensive disorder of pregnancy diagnosed antepartum or intrapartum

requiring blood pressure medication in the postpartum

Chronic hypertension requiring blood pressure medication postpartum

**Exclusion Criteria** 

Urine output < 30 cc/h prior to screening for eligibility</li>

IRB NUMBER: HSC-MS-21-0476 UTHealth IRB APPROVAL DATE: 07/06/2022

Creatinine > 1.4 during current admission

End-stage renal disease

Hypersensitivity to ACE inhibitors or sulfa drugs

Idiopathic/hereditary angioedema

Hyperkalemia (serum potassium >5 mEq/L) during current admission

Pulmonary edema

Randomization:

Randomization will be achieved by computer-generated random sequences that

will be created by a non-clinical member of the research team. A permuted block

randomization with a random fashion will be used to prevent imbalances between

groups.

Randomization will be stratified according to:

1. Primary diagnosis: chronic hypertension or newly diagnosed preeclampsia

2. Recruiting site

Setting:

Recruitment will occur on the Labor and Delivery ward and postpartum ward at:

Memorial Hermann Hospital-Sowthwest.

Lyndon B. Johnson Hospital

Memorial Hermann Hospital-Texas Medical Center.

Recruitment

The research staff/MFM physician will approach individuals that meet the

inclusion and exclusion criteria during their hospital stay before discharge.

The research stuff will Introduce Babyscripts as a health system's mobile app

and sign the patients up for Babyscripts.

After adding the patient to the system, the patient will receive an email and a text

message with a personal passcode to complete registration.

The patient will download the Babyscripts myJourney app on her smartphone

and enter the personal passcode under "New User" where it indicates. From

there, the patient will be prompted to fill in some additional information to

complete registration.

o Once the patient completes registration, we will provide her with a BP monitor so

you can start taking readings through the app.

The patients will be instructed to monitor their BP twice daily, in the morning and

the evening.

Of Note, Babyscripts sends daily SMS reminders, twice a day, to remind patients

to check their blood pressure.

Intervention and procedures

Participants will be randomized to Hctz/Lisinopril (brand name: Zestoretic) or

extended release Nifedipine. Group 1 will be composed of women allocated to

Hctz/Lisinopril treatment. Group 2 will be composed of women allocated to

extended release Nifedipine treatment.

Hctz/Lisinopril and extended release Nifedipine will be administrated orally in the

morning for both groups.

The allocated study medication will be incrementally increased to achieve blood

pressure control according to the threshold listed below (Table 2).

- If maximum dose of one medication will be reached without blood pressure control, oral labetalol will be added at the lowest dose increasing as needed.
- Hctz/Lisinopril will be started at 10mg/12.5 daily
- Extended release Nifedipine will be starts at 30mg daily
- The use of concomitant intravenous antihypertensive medication (i.e. Hydralazine, labetalol) for severe hypertension as well as the use of magnesium sulfate for seizure prophylaxis will be left to the discretion of the treating medical team
- Following hospital discharge, twice a day (8am and 7pm), patients will receive SMS and push notifications to remind them to take their BP through the Babyscript app. If patients have three missed readings in a row, they will receive a SMS and push notification.
- o information will be collected from the medical record including medical and pregnancy history, lab results, delivery and postpartum information.

Table 2: Dose adjustment plan

| | Initial | Dosing adjustment | Maximum |
|--------------------------------|---------|-------------------|-----------|
| | dose | | dose/day |
| Extended release Nifedipine | 30mg/ | Increase by | 90mg/day |
| | day | 30mg/day | |
| Lisinopril/Hydrochlorothiazide | 10mg/ | Increase by 10mg | 20/25/day |
| | 12.5m | lisinopril/day to | |
| | g/day | 20mg/12.5 mg | |

| Next increase will be |
|-----------------------|
| with the HCTZ to |
| 20mg/25 |

Thresholds for action based on raised blood pressure in the postpartum period:

The following recommendations for blood pressure treatment in the postpartum period are based on the ACOG and NICE guidelines<sup>38</sup>

## During hospital stay:

- o SBP≥160 or DBP≥110, repeat BP in 15 minutes
- If persistent, give intravenous medication to lower blood pressure and increase oral medication the next morning
- SBP ≥150 or DBP≥100, repeat BP in 4 hours
- If persistent, increase oral medication the next morning

### After discharge from the hospital

- SBP≥160 or DBP≥110, repeat BP in 15 minutes
- o If persistent, refer for evaluation in the clinic or the emergency department
- SBP≥150 or DBP≥100 in BP monitoring at home or in postpartum clinic,
   increase oral medication the next morning

#### Outcome measures:

- All patients will receive a Bluetooth BP cuff at during the hospital course.
- The BP cuff will be connected via Bluetooth to a Babyscripts application and available for the research team to review (Figure 1).

 The Babyscripts app is a resource for all UT Physicians obstetrical patients during their pregnancy and postpartum.

 The participants will be instructed to measure their BP twice daily until their clinic appointment.

 Following their postpartum clinic appointment the participants will be instructed to measure their BP once daily.

 All patients will be followed in the clinic 7-10 days after delivery and 6 weeks postpartum as recommended by the ACOG guidelines

Patients will be contacted 3 month, 6 month and 1 year after delivery by
 telephone for information regarding blood pressure control, medication use.

Figure:



# Primary outcome:

Stage 2 hypertension at day 7-10 after delivery (defined as SBP ≥ 140 and/or DBP ≥ 90 mmHg) or admission to the hospital for blood pressure control prior to day 10.

Primary outcome will be calculated as the average BP reading for day 7-10 after delivery.

# Secondary outcomes:

- Occurrence of severe postpartum hypertension (SBP≥160 and/or DBP≥110 mmHg on 2 occasions, 15 minutes apart)
- Receipt of additional antihypertensive during admission, at 7-10 postpartum, and at 6 weeks postpartum.

- Postpartum length of stay
- Postpartum readmission
- Time from delivery to BP control (i.e time from delivery to last BP <150/100).
- Incidence of persistent postpartum hypertension 6 weeks postpartum (SBP ≥ 140 and/or DBP ≥ 90 mmHg).
- Proteinuria at 7-10 days, and 6 weeks postpartum (measured by urine protein creatinine ratio).
- Labs abnormality including hyperkalemia or creatinine increase at 7-10 day visit and 6 weeks postpartum.
- Compliance with medications at postpartum visit at 7-10 days after delivery and 6
  weeks postpartum. The patient will be asked to bring their medication bottle with
  them and the compliance will be measured by counting pills at each postpartum
  visit.
- Blood pressure control at 3 month, 6 month, 9 month, 1 year after delivery and need for BP medications.
- % of patients receiving primary care with BP measurement at 1 year.
- Postpartum complications captured as Severe composite maternal morbidity:
  - Need for ICU admission
  - HELLP
  - Eclampsia
  - Stroke
  - Renal failure
  - Pulmonary edema

Cardiomyopathy

Maternal death

Blood pressure control at 3 month, 6 month, 9 month, 1 year after delivery and

need for BP medications

• % of patients receiving primary care with BP measurement at 1 year

Sample size:

Due to lack of information regarding the prevalence of persistent hypertension 7 days

after delivery, and the limited information regarding the use of ACE inhibitors in the

postpartum period, this will be a pilot study that will include 70 patients. That sample

size will allow us to gather information regarding feasibility, compliance, rate of the

primary outcome, dosing of medications, and side effects.

Feasibility:

Based on data from our center, in the 3 participating centers there are 6,574 deliveries

per year. With 10% rate of preeclampsia, 657 people per year will be eligible to

participate in this trial. Assuming 30-50% of patients will decline to participate, we will

expect to recruit 70 patients in 6-9 month.

Blinding:

We will not be able to blind the treating physician or patient to the study

medication due to different dose adjustment, side effects, etc.

However, the research person who would review the 7-10 day BP measurements

will be blinded to treatment assignment

**Procedures for safety monitoring:** 

UTHealth
The University of Texas
Health Science Center at Houston

A review of the available observational literature concluded that extended release

nifedipine and ACEI have minimal milk to maternal plasma ratios to make

breastfeeding acceptable.

Additionally Severe BP (SBP≥160/DBP ≥110) will be reported by the babyscript

app to the physician via text and email, and the team will contact the patient for

further management

Statistical tests:

An intent-to-treat analysis will be conducted. Outcomes will be evaluated using

the independent t-test for continuous variables and the x<sup>2</sup> or fisher's exact test for

categorical variables as appropriate. Mann-Whitney U test will be used for non-

parametric comparisons. We will report RR and 95% confidence intervals.

Secondary outcome measures will be compared.

We will conduct a Bayesian analysis to calculate the probability of treatment

benefit or hram. The probability of at least 20% reduction in the rate of the

primary outcome will be considered clinically significant, we conservatively set a

neutral prior probability centered at a relative risk (RR) of 1.0 (i.e., a priori no

effect on the outcome) and a 95% credible interval of 0.25 - 4.0.

**Ancillary Studies** 

1. Medication adherence survey: Medication non- adherence is an important public

health issue that clinicians encounter. Approximately 78% of e-prescriptions are

actually filled; only 72% of new prescriptions are filled. 48 Non-compliance is most common among new prescriptions for chronic conditions including hypertension(31.4%). Adherence to medications can be affected by a variety of factors in patients with hypertension; the perception that drugs are only needed when blood pressure levels are high, concerns regarding adverse effects, and lack of self-confidence in their self-treatment. Medications are commonly used in pregnancy and postpartum, with at least 81.2-96.9% of women using at least one medication, either prescribed or over-the-counter. 49,50 The attitudes regarding drug use in pregnancy and obtaining drug information play an essential role in medication adherence<sup>51</sup>. The MMAS-8 validated survey (attached as Figure 1) will be given to women to complete their routine postpartum care during their clinic visit if they meet study criteria and agree to the study. This survey will be supplemented with other questions about demographics and challenges with prescription error and pick-up problems. It takes less than 10 minutes to complete. The answers will not be available to the managing health care provider but will be kept in the locked research office until after the delivery of the subject. Based on the survey scores, the subject will be divided into groups based on high, medium and low adherence. Outcomes between groups will be compared.

2. Social determinants of health (SDH) Survey (SDH)- while our approach to clinical care is rooted in biology, an increasingly interdisciplinary approach is being employed that acknowledges SDH, i.e., the social and structural aspects of a 'patient's life that can influence health. Social determinants of health (SDH) include but are not limited to basic resources, educational opportunities and economic stability, access to health care,

community resources, literacy, socioeconomics, and safety. 52 By understanding SDH, interventions can be pursued that can improve individual and population health. For patients living with hypertension, there is a correlation between social determinants of health and blood pressure control. SDH also impacts many obstetrical conditions. 53 Using this broader context to understand 'patients' health care decision-making and health literacy facilitates the intersections of social identity and their associated patterns of structural oppression and fosters a creative approach to overcoming potential barriers. The PRAPARE Assessment (The Protocol for Responding to and Assessing' Patients' Assets, Risks, and Experiences) is an established tool to assess SDH briefly. Core measures of this tool include race, ethnicity, education, employment, insurance, income, material security, transportation, social integration and support, stress and migrant, veteran and housing status. It will provide insight by which we can understand correlations between SDH and health care outcomes in our population as a springboard to improving both the outcomes and the pathways leading to them. The brevity of questions covering numerous social domains can help target particular social features that may be correlated with blood pressure control as well as target resource referrals and utilization, thereby translating into actionable items.

### **Ethical considerations**

### Informed consent

All study candidates will be given a full explanation of study, allowed to read the informed consent, and be provided the opportunity to ask any questions. Once all questions have been answered and the investigator is assured that the individual



understands the requirements of the study, the subject will be signing an informed

consent. The investigator shall provide a copy of the informed consent.

Institutional review board

Before initiation of the study, the PI will obtain approval of the research protocol from

the IRB. The study will be registered in www.clinicaltrials.gov as required by US law for

public access.

Subject confidentially

Each study's subject anonymity will be maintained throughout the study. Before

collecting the data, a unique study number will be assigned to each case, thus de-

identifying the individual subject. There will be a log of the study subject to the assigned

study number in the study site.

Research assistants are in compliance with required CITI training. When the results of

this research study are reported in medical journals or at scientific meetings, the

subjects who take part will not be named or identified. The Federal Privacy Act protects

the confidentiality of medical records and any private health information collected.

Access to personal data will be limited to the investigators only. However, these

individuals are required to keep all information confidential.

Data handling and record-keeping

Access to source documents:

UTHealth
The University of Texas
Health Science Center at Houston

IRB NUMBER: HSC-MS-21-0476
THealth IRB APPROVAL DATE: 07/06/2022

Research personal will perform data collection manually from patient charts at the

different sites. Please refer to the attached data collection sheet for detail on variables

to be collected. Data will be collected from randomization until one year postpartum.

Records retention: Data will be digitally encrypted and stored in the UTHealth Redcap

system. After the study, the principal investigator will retain copies of the approved

protocol and all other supporting documentation related to the project. De-identified

patient information may be used for future research projects.

Quality control Assurance: the principal investigator and co-investigators will go

through all the files to assure that data is reliable and complete. The verification will be

by self-assessment.

Figure 1: Morisky Medication Adherence Questions (MMAS-8).

These are questions about your medication adherence. Please circle or select one

option.

1. Do you sometimes forget to take your medicine?

No Yes

2. People sometimes miss taking their medicines

No Yes



for reasons other than forgetting. Were there any days when you did not take your medicine?

- 3. Have you ever cut back or stopped taking your No Yes medicine without telling your doctor because you felt worse when you took it?
- 4. When you travel or leave home, do you sometimes No Yes forget to bring along your medicine?
- 5. Did you take all your medicines yesterday? No Yes
- 6. When you feel like your symptoms are under control, No Yes do you sometimes stop taking your medicine?
- 7. Taking medicine every day is a real inconvenience No Yes for some people. Do you ever feel hassled about sticking to your treatment plan?

| 8. How often do you have difficulty remembering to |
|----------------------------------------------------|
| take all your blood pressure medication? |
| A. Never/rarely |
| B. Once in a while |
| C. Sometimes |
| D. Usually |
| E. All the time |

### References:

- 1. Umesawa M, Kobashi G. Epidemiology of hypertensive disorders in pregnancy: prevalence, risk factors, predictors and prognosis. Hypertens Res. 2017;40(3):213-220.
- 2. Murray Horwitz ME, Rodriguez MI, Dissanayake M, Carmichael SL, Snowden JM. Postpartum health risks among women with hypertensive disorders of pregnancy, California 2008-2012. J Hypertens. 2020.
- 3. Too G, Wen T, Boehme AK, et al. Timing and Risk Factors of Postpartum Stroke. Obstet Gynecol. 2018;131(1):70-78.
- Evans CS, Gooch L, Flotta D, et al. Cardiovascular system during the postpartum 4. state in women with a history of preeclampsia. *Hypertension*. 2011;58(1):57-62.
- Melchiorre K, Sutherland GR, Liberati M, Thilaganathan B. Preeclampsia is 5. associated with persistent postpartum cardiovascular impairment. Hypertension. 2011;58(4):709-715.
- Arnott C, Nelson M, Alfaro Ramirez M, et al. Maternal cardiovascular risk after 6. hypertensive disorder of pregnancy. Heart. 2020;106(24):1927-1933.
- 7. Grandi SM, Filion KB, Yoon S, et al. Cardiovascular Disease-Related Morbidity and Mortality in Women With a History of Pregnancy Complications. Circulation. 2019;139(8):1069-1079.
- 8. Leon LJ, McCarthy FP, Direk K, et al. Preeclampsia and Cardiovascular Disease in a Large UK Pregnancy Cohort of Linked Electronic Health Records: A CALIBER Study. Circulation. 2019;140(13):1050-1060.



- 9. Lykke JA, Langhoff-Roos J, Sibai BM, Funai EF, Triche EW, Paidas MJ. Hypertensive pregnancy disorders and subsequent cardiovascular morbidity and type 2 diabetes mellitus in the mother. Hypertension. 2009;53(6):944-951.
- 10. McDonald SD, Malinowski A, Zhou Q, Yusuf S, Devereaux PJ. Cardiovascular sequelae of preeclampsia/eclampsia: a systematic review and meta-analyses. Am Heart J. 2008;156(5):918-930.
- 11. Wikstrom AK, Haglund B, Olovsson M, Lindeberg SN. The risk of maternal ischaemic heart disease after gestational hypertensive disease. BJOG. 2005;112(11):1486-1491.
- 12. Giorgione V, Ridder A, Kalafat E, Khalil A, Thilaganathan B. Incidence of postpartum hypertension within 2 years of a pregnancy complicated by preeclampsia: a systematic review and meta-analysis. *BJOG.* 2020.
- 13. Bellamy L, Casas JP, Hingorani AD, Williams DJ. Preeclampsia and risk of cardiovascular disease and cancer in later life: systematic review and metaanalysis. BMJ. 2007;335(7627):974.
- 14. American College of O, Gynecologists, Task Force on Hypertension in P. Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013;122(5):1122-1131.
- 15. Blue NR, Murray-Krezan C, Drake-Lavelle S, et al. effect of ibuprofen vs acetaminophen on postpartum hypertension in preeclampsia with severe features: a double-masked, randomized controlled trial. Am J Obstet Gynecol. 2018;218(6):616 e611-616 e618.
- Goel A, Maski MR, Bajracharya S, et al. Epidemiology and Mechanisms of De 16. Novo and Persistent Hypertension in the Postpartum Period. *Circulation*. 2015;132(18):1726-1733.
- 17. Berks D, Steegers EAP, Molas M, Visser W. Resolution of hypertension and proteinuria after preeclampsia. Obstet Gynecol. 2009;114(6):1307-1314.
- Cairns AE, Pealing L, Duffy JMN, et al. Postpartum management of hypertensive 18. disorders of pregnancy: a systematic review. BMJ Open. 2017;7(11):e018696.
- 19. Hirshberg A, Levine LD, Srinivas SK. Clinical factors associated with readmission for postpartum hypertension in women with pregnancy-related hypertension: a nested case control study. J Perinatol. 2016;36(5):405-409.
- Matthys LA, Coppage KH, Lambers DS, Barton JR, Sibai BM. Delayed 20. postpartum preeclampsia: an experience of 151 cases. Am J Obstet Gynecol. 2004;190(5):1464-1466.
- 21. Barton JR, Hiett AK, Conover WB. The use of nifedipine during the postpartum period in patients with severe preeclampsia. Am J Obstet Gynecol. 1990;162(3):788-792.
- 22. Vermillion ST, Scardo JA, Newman RB, Chauhan SP. A randomized, doubleblind trial of oral nifedipine and intravenous labetalol in hypertensive emergencies of pregnancy. Am J Obstet Gynecol. 1999;181(4):858-861.
- Arias-Hernandez G, Vargas-De-Leon C, Calzada-Mendoza CC, Ocharan-23. Hernandez ME. Efficacy of Diltiazem for the Control of Blood Pressure in Puerperal Patients with Severe Preeclampsia: A Randomized, Single-Blind, Controlled Trial. Int J Hypertens. 2020;2020:5347918.



- 24. Fidler J, Smith V, De Swiet M. A randomized study comparing timolol and methyldopa in hospital treatment of puerperal hypertension. *Br J Obstet Gynaecol.* 1982;89(12):1031-1034.
- 25. Mabie WC, Gonzalez AR, Sibai BM, Amon E. A comparative trial of labetalol and hydralazine in the acute management of severe hypertension complicating pregnancy. *Obstet Gynecol.* 1987;70(3 Pt 1):328-333.
- 26. Sharma KJ, Greene N, Kilpatrick SJ. Oral labetalol compared to oral nifedipine for postpartum hypertension: A randomized controlled trial. *Hypertens Pregnancy*. 2017;36(1):44-47.
- 27. Matthews G, Gornall R, Saunders NJ. A randomised placebo controlled trial of loop diuretics in moderate/severe preeclampsia, following delivery. *J Obstet Gynaecol.* 1997;17(1):30-32.
- 28. Ascarelli MH, Johnson V, McCreary H, Cushman J, May WL, Martin JN, Jr. Postpartum preeclampsia management with furosemide: a randomized clinical trial. *Obstet Gynecol.* 2005;105(1):29-33.
- 29. Veena P, Perivela L, Raghavan SS. Furosemide in postpartum management of severe preeclampsia: A randomized controlled trial. *Hypertens Pregnancy*. 2017;36(1):84-89.
- 30. Viteri OA, Alrais MA, Pedroza C, et al. Torsemide for Prevention of Persistent Postpartum Hypertension in Women With Preeclampsia: A Randomized Controlled Trial. *Obstet Gynecol.* 2018;132(5):1185-1191.
- 31. Lopes Perdigao J, Lewey J, Hirshberg A, et al. Furosemide for Accelerated Recovery of Blood Pressure Postpartum in women with a hypertensive disorder of pregnancy: A Randomized Controlled Trial. *Hypertension*. 2021:HYPERTENSIONAHA12016133.
- 32. Ormesher L, Higson S, Luckie M, et al. Postnatal Enalapril to Improve Cardiovascular Function Following Preterm Preeclampsia (PICk-UP):: A Randomized Double-Blind Placebo-Controlled Feasibility Trial. *Hypertension*. 2020;76(6):1828-1837.
- 33. Noronha Neto C C, Maia SS, Katz L, Coutinho IC, Souza AR, Amorim MM. Clonidine versus Captopril for Severe Postpartum Hypertension: A Randomized Controlled Trial. *PLoS One.* 2017;12(1):e0168124.
- 34. Griffis KR, Jr., Martin JN, Jr., Palmer SM, Martin RW, Morrison JC. Utilization of hydralazine or alpha-methyldopa for the management of early puerperal hypertension. *Am J Perinatol.* 1989;6(4):437-441.
- 35. Vigil-De Gracia P, Ruiz E, Lopez JC, de Jaramillo IA, Vega-Maleck JC, Pinzon J. Management of severe hypertension in the postpartum period with intravenous hydralazine or labetalol: a randomized clinical trial. *Hypertens Pregnancy*. 2007;26(2):163-171.
- 36. Beardmore KS, Morris JM, Gallery ED. Excretion of antihypertensive medication into human breast milk: a systematic review. *Hypertens Pregnancy*. 2002;21(1):85-95.
- 37. Sibai BM. Etiology and management of postpartum hypertension-preeclampsia. *Am J Obstet Gynecol.* 2012;206(6):470-475.
- 38. In: *Hypertension in pregnancy: diagnosis and management.* London2019.



- 39. Podymow T. Joseph G. Preconception and pregnancy management of women with diabetic nephropathy on angiotensin converting enzyme inhibitors. Clin Nephrol. 2015;83(2):73-79.
- 40. Heart Outcomes Prevention Evaluation Study I, Yusuf S, Sleight P, et al. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. N Engl J Med. 2000;342(3):145-153.
- 41. Magee L, von Dadelszen P. Prevention and treatment of postpartum hypertension. Cochrane Database Syst Rev. 2013(4):CD004351.
- 42. Redman CW, Kelly JG, Cooper WD. The excretion of enalapril and enalaprilatin human breast milk. Eur J Clin Pharmacol. 1990;38(1):99.
- 43. Bramham K, Nelson-Piercy C, Brown MJ, Chappell LC. Postpartum management of hypertension. BMJ. 2013;346:f894.
- 44. Shannon ME, Malecha SE, Cha AJ. Angiotensin converting enzyme inhibitors (ACEIs) and angiotensin II receptor blockers (ARBs) and lactation: an update. J Hum Lact. 2000;16(2):152-155.
- 45. Chesley LC. Vascular reactivity in normal and toxemic pregnancy. *Clin Obstet* Gynecol. 1966;9(4):871-881.
- Gant NF, Daley GL, Chand S, Whalley PJ, MacDonald PC. A study of 46. angiotensin II pressor response throughout primigravid pregnancy. J Clin Invest. 1973;52(11):2682-2689.
- 47. Saxena AR, Karumanchi SA, Brown NJ, Royle CM, McElrath TF, Seely EW. Increased sensitivity to angiotensin II is present postpartum in women with a history of hypertensive pregnancy. Hypertension. 2010;55(5):1239-1245.
- 48. Fischer MA, Stedman MR, Lii J, et al. Primary medication non-adherence: analysis of 195,930 electronic prescriptions. J Gen Intern Med. 2010;25(4):284-290.
- 49. Lupattelli A, Spigset O, Nordeng H. Adherence to medication for chronic disorders during pregnancy: results from a multinational study. Int J Clin Pharm. 2014;36(1):145-153.
- 50. Refuerzo JS, Blackwell SC, Sokol RJ, et al. use of over-the-counter medications and herbal remedies in pregnancy. Am J Perinatol. 2005;22(6):321-324.
- Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-51. reported measure of medication adherence. Med Care. 1986;24(1):67-74.
- 52. Braveman P, Gottlieb L. The social determinants of health: it's time to consider the causes of the causes. Public Health Rep. 2014;129 Suppl 2:19-31.
- 53. Committee on Health Care for Underserved W. ACOG Committee Opinion No. 729: Importance of Social Determinants of Health and Cultural Awareness in the Delivery of Reproductive Health Care. Obstet Gynecol. 2018;131(1):e43-e48.